CLINICAL TRIAL: NCT04686994
Title: A Randomized, Double-Blind, Placebo-Controlled Phase Ib Study to Evaluate Safety, Tolerability and Pharmacokinetics and Pharmacodynamics (Biomarkers) of ASC41 Tables in Overweight and Obese Subjects
Brief Title: Study to Evaluate the Safety and Efficacy of ASC41 in Overweight and Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Collaborators: Hunan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASC41-104
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Overweight and Obesity; NAFLD; Hyperlipidemia
Keywords: Overweight and Obesity; NAFLD; Hyperlipidemia; LDL-C; NASH
MeSH Terms: conditions — Overweight; Obesity; Non-alcoholic Fatty Liver Disease; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Parallel Assignment 3:1 ratio
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASC41 (Experimental): ASC41 two tablets, once daily, from Day 1 to Day 28.
  Interventions: Drug: ASC 41
- ASC41 placebo (Placebo Comparator): ASC41 placebo two tablets, once daily, from Day 1 to Day 28.
  Interventions: Drug: ASC 41 Placebo

INTERVENTIONS:
Drug: ASC 41 — Oral tablets
  Arms: ASC41
Drug: ASC 41 Placebo — Oral tablets
  Arms: ASC41 placebo

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability and compare the pharmacokinetic parameters of ASC41, a THR beta agonist tables in overweight and obese subjects who have elevated LDL-C .

ELIGIBILITY:
Key Inclusion Criteria:

* 23kg/m2 ≤ BMI <40kg/m2.

Key Exclusion Criteria:

* A history of thyroid disease.
* A positive HBsAg, HCV Ab and/or HIV Ab.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-02-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 28 days
  Occurrence of Serious Adverse Event (SAE), Adverse Event (AE) resulting in treatment discontinuation and/or dose reductions, and AE of special interest, from baseline up to 28 days

SECONDARY OUTCOMES:
AUC of ASC41 | Up to 28 days
  Evaluate the Area under the plasma concentration versus time curve after multiple oral doses of ASC41 tablets.
Cmax of ASC41 | Up to 28 days
  Evaluate the Peak Plasma Concentration after single and multiple oral doses of ASC41 tablets.
t1/2 of ASC41 | Up to 28 days
  Evaluate the Terminal-Phase Half-Life after single and multiple oral doses of ASC41 tables.
CL/F of ASC41 | Up to 28 days
  Evaluate the Apparent Systemic Clearance after multiple oral dose of ASC41 tables.
Vd/F of ASC41 | Up to 28 days
  Evaluate the Apparent Systemic Clearance after multiple oral dose of ASC41 tables.
Tmax of ASC41 | Up to 28 days
  Evaluate the Time to reach the maximum plasma concentration after multiple oral doses of ASC41 tables.
LDL-C and other lipid parameters | Up to 28 days
  To evaluate the effect of multiple doses of ASC41 tablets on LDL-C and other lipid parameters (TG, TC, HDL-C, etc.) .

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan provincial people's hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided